CLINICAL TRIAL: NCT06515561
Title: Prevalence of Teeth Discoloration and Associated Risk Factors and Determination of the Most Common Shade Among Group of Egyptian Population: Educational Hospital Based Cross Sectional Study
Brief Title: Prevalence of Teeth Discoloration , Associated Risk Factors and the Most Common Shade Among Group of Egyptian Population
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Mohamed Saber Abd Al Aziz, assistant lecturer at conservative department, Cairo University
Other Study IDs: PREVELANCE OF DISCOLORATION
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Discoloration, Tooth
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
"The aim of this study is to assess the prevalence of tooth discoloration and explore its associated risk factors, including local cultural practices or environmental conditions, among a group of adults aged 20 to 45 years in an Egyptian population sample. Moreover, we aim to identify the most common dental shades in the same sample."

DETAILED DESCRIPTION:
Discoloration of teeth is a frequent dental finding and it is often esthetically displeasing and psychologically traumatizing to the patient (Manuel et al., 2010). Changes in the three distinct layers of the tooth; enamel, dentin and cementum are known to cause modification in the appearance of the teeth leading to a change in its light transmission and reflection properties (Watts et al., 2001). Generally, tooth discoloration is said to have occurred when there is a deviation in tooth color. Suresh and Gopi in 2010 noted that the normal color of primary teeth is bluish white, whereas the color of permanent teeth is grayish white or yellowish white. The teeth of adults usually appear more yellow or grayish yellow than those of younger persons because as one ages, the enamel becomes thinner from physiological wear, while the dentin becomes thicker from the deposition of secondary dentin. There are two types of tooth discoloration, extrinsic and intrinsic, while the extrinsic type is apparent on the outer surface of the teeth, the intrinsic type stains are coming from inside of the teeth. The main cause of intrinsic tooth discoloration is the decomposition of pulp tissue, which is the first indication of pulp death (Suresh & Gopi., 2010). Other causes of intrinsic tooth discoloration are enamel opacities, dental caries, tetracycline, minocycline and doxycycline staining, and enamel hypoplasia (Koleoso et al., 2004). These medications can leave a characteristic bright-yellow band that fluoresces under ultraviolet light (tetracycline) or a green-gray or blue-gray intrinsic staining (minocycline). Also, Fluoride can cause enamel discoloration through hypomineralization when too much of it is ingested during the early maturation stage of enamel formation. In addition, dental materials used for dental restorations like amalgam restorations, can generate corrosion products such as silver sulfide which can leave a gray-black color on the teeth.

On the other hand, extrinsic dental discoloration might be due to tea, coffee, tobacco smoking/chewing, betel nut chewing, drugs (e.g., chlorhexidine mouth rinse), iron salts, heavy metals (e.g., silver nitrate and lead), essential oils, amoxicillin-clavulinic acid, ciprofloxacin, linezolide, and glibenclamide (Kumar et al., 2012). Enamel defects, salivary dysfunction, and poor oral hygiene could be predisposing factors to extrinsic discoloration. Small pits and defects on the outer surface of the enamel can lead to an accumulation of food particles and stains from beverages, tobacco, and other topical agents on its surface causing the discoloration. Salivary dysfunction such as, decreased salivation can lead to difficulties in removing food debris from the tooth surface and can thus contribute to the staining of teeth. Conditions that are associated with a reduction in the salivation are salivary gland obstruction and infection, Sjögren syndrome, head and neck radiation therapy for cancer, chemotherapy, and multiple medications (e.g., anticholinergics, antihypertensive, antipsychotics and antihistamines). All of these can cause teeth discoloration (Patel et al., 2013).

ELIGIBILITY:
Inclusion Criteria:

* Age 20-45 years.
* Males or females.
* Egyptians.
* Presence of at least 20 teeth in function.
* Patient compliance.

Exclusion Criteria:

* Psychologically unstable or mentally retarded participants
* Participants with severe periodontal diseases.
* Participants in need for emergency intervention

Ages: 20 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Egyptian adults of both sexes aged 20-45 years from outpatient clinic, Faculty of Dentistry, Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
prevalence and severity of discoloration | 3 months
  assessment of the prevalence and severity of dental discoloration among adults in the study area.

SECONDARY OUTCOMES:
risk factors and their association with discoloration | 3 months
  Identification of risk factors and their association with discoloration in the study population and knowing the most common teeth shade among the same group of population.
Most common teeth shade | 3 months
  determination of most common teeth shade usingVita classical shade guide

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Yassen, ph degree, Study Director — Professor at Conservative Dentistry Department, Faculty of Dentistry, Cairo University.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Koleoso DC, Shaba OP, Isiekwe MC. Prevalence of intrinsic tooth discolouration among 11-16 year-old Nigerians. Odontostomatol Trop. 2004 Jun;27(106):35-9. PMID 15536720